CLINICAL TRIAL: NCT00972374
Title: Safety and Efficacy of Brimonidine Tartrate Posterior Segment Drug Delivery System in Improving Visual Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 190342-031D
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Results first posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-03

CONDITIONS: Rhegmatogenous Macula-off Retinal Detachment
MeSH Terms: interventions — Brimonidine Tartrate; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 400 ug Brimonidine Implant (Experimental): 400 ug Brimonidine Tartrate Posterior Segment Drug Delivery system on Day 1 in the study eye.
  Interventions: Drug: 400 ug Brimonidine Implant
- 200 ug Brimonidine Implant (Experimental): 200 ug Brimonidine Tartrate Posterior Segment Drug Delivery system on Day 1 in the study eye.
  Interventions: Drug: 200 ug Brimonidine Implant
- Sham (no implant) (Sham Comparator): Sham Posterior Segment Drug Delivery system on Day 1 in the study eye.
  Interventions: Other: Sham (no implant)

INTERVENTIONS:
Drug: 400 ug Brimonidine Implant — 400 ug Brimonidine Tartrate Posterior Segment Drug Delivery system on Day 1 in the study eye.
  Other Names: Brimonidine Tartrate PS DDS®
  Arms: 400 ug Brimonidine Implant
Drug: 200 ug Brimonidine Implant — 200 ug Brimonidine Tartrate Posterior Segment Drug Delivery system on Day 1 in the study eye.
  Other Names: Brimonidine Tartrate PS DDS®
  Arms: 200 ug Brimonidine Implant
Other: Sham (no implant) — Sham Posterior Segment Drug Delivery system on Day 1 in the study eye.
  Arms: Sham (no implant)

SUMMARY:
This study will evaluate the efficacy and safety of the Brimo PS DDS® Applicator System (200 μg and 400 μg brimonidine tartrate) on visual function in patients with previous rhegmatogenous macula-off retinal detachment.

ELIGIBILITY:
Inclusion Criteria:

* The macula-off retinal detachment must have been caused by a rupture (rhegmatogenous in etiology)
* The repair of the macula-off retinal detachment must have occurred at least 6 months before the Day 1 visit in the study eye
* The repair must have been deemed an anatomic success and required no more than one macular re-attachment procedure
* The visual acuity score must be between 20/50 and 20/320 in the study eye

Exclusion Criteria:

* Any sight-threatening ocular condition in the study eye other than the ruptured retinal detachment
* Anticipated need for ocular surgery during the 12-month study period
* Any injectable, periocular, or intravitreal corticosteroid treatment to study eye within 6 months prior to screening (eg, triamcinolone acetonide)
* Any injectable, periocular, or intravitreal anti-VEGF treatment to the study eye within 3 months prior to screening (eg, Avastin or Lucentis)
* Any infectious condition in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (6):
- Abilene, Texas, United States
- New Delhi, India
- Tel Aviv, Israel
- Makati, Philippines
- Seoul, South Korea
- London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 400 ug Brimonidine Implant | 200 ug Brimonidine Implant | Sham (no Implant)
Started | 15 | 15 | 14
Completed | 13 | 15 | 13
Not Completed | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 400 ug Brimonidine Implant | 200 ug Brimonidine Implant | Sham (no Implant) | Total
Number analyzed (Participants) | 15 | 15 | 14 | 44
Age Continuous [Mean (Standard Deviation); unit: Years] | 54.2 (17.12) | 54.3 (20.36) | 56.1 (15.19) | 54.9 (17.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 5 | 16
  Male | 9 | 10 | 9 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With at Least a 15-Letter Increase From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly indicates that vision has improved. The percentage of patients with at least a 15-letter increase in BCVA in the study eye is reported.
Time Frame: Month 3
Population: Intent to Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | 400 ug Brimonidine Implant | 200 ug Brimonidine Implant | Sham (no Implant)
Number analyzed (Participants) | 15 | 15 | 14
Percentage of Patients | 6.7 | 6.7 | 0

2. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening.
Time Frame: Baseline, Month 3
Population: Intent to Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Number of Letters Read Correctly
Arm/Group | 400 ug Brimonidine Implant | 200 ug Brimonidine Implant | Sham (no Implant)
Number analyzed (Participants) | 15 | 15 | 14
Number of Letters Read Correctly
  Baseline | 46.6 (13.69) | 53.3 (8.46) | 50.3 (10.92)
  Change from Baseline at Month 3 | 6.0 (6.23) | 3.1 (6.78) | 4.8 (4.64)

3. Other Pre Specified Outcome: Percentage of Patients With Intraocular Pressure (IOP) < 10 mmHg in the Study Eye at Any Follow up Visit
Description: IOP is the fluid pressure inside the eye. The percentage of patients with IOP < 10 millimeters of mercury (mmHg) in the study eye at any follow up visit is presented.
Time Frame: 12 Months
Population: Intent to Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | 400 ug Brimonidine Implant | 200 ug Brimonidine Implant | Sham (no Implant)
Number analyzed (Participants) | 15 | 15 | 14
Percentage of Patients | 20.0 | 26.7 | 28.6

ADVERSE EVENTS:
Description: For Ocular Adverse Events (AEs), only those in the study eye are reported in the "Other Adverse Events" section. For Serious Adverse Events (SAEs), all ocular events are reported in the SAE section, regardless of the eye.
Arm/Group | 400 ug Brimonidine Implant | 200 ug Brimonidine Implant | Sham (no Implant)
Serious Adverse Events (participants affected / at risk) | 0/15 | 2/15 | 2/14
Other Adverse Events (participants affected / at risk) | 7/15 | 12/15 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 400 ug Brimonidine Implant (N=15) | 200 ug Brimonidine Implant (N=15) | Sham (no Implant) (N=14)
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Prostate Cancer [y] (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9 | 1/10 | 0/9
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Strabismus Correction (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 400 ug Brimonidine Implant (N=15) | 200 ug Brimonidine Implant (N=15) | Sham (no Implant) (N=14)
Conjunctival Haemorrhage (Eye disorders) | 3 | 1 | 2
Conjunctival Hyperaemia (Eye disorders) | 2 | 1 | 1
Eye Pruritus (Eye disorders) | 2 | 0 | 0
Eye Pain (Eye disorders) | 1 | 3 | 1
Hypotony of Eye (Eye disorders) | 1 | 2 | 0
Intraocular Pressure Decreased (Investigations) | 1 | 2 | 0
Conjunctival Oedema (Eye disorders) | 1 | 1 | 1
Maculopathy (Eye disorders) | 1 | 1 | 0
Cataract Subscapular (Eye disorders) | 1 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0
Retinal Haemorrhage (Eye disorders) | 1 | 0 | 1
Vitreous Floaters (Eye disorders) | 1 | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 0
Cataract Nuclear (Eye disorders) | 1 | 0 | 0
Eye Irritation (Eye disorders) | 1 | 0 | 0
Influenza Like Illness (General disorders) | 1 | 0 | 0
Keratoconjunctivitis Sicca (Eye disorders) | 1 | 0 | 0
Optic Atrophy (Eye disorders) | 1 | 0 | 0
Optic Disc Haemorrhage (Eye disorders) | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Vitreous Haemorrhage (Eye disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0
Posterior Capsule Opacification (Eye disorders) | 0 | 1 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 1
Anterior Chamber Inflammation (Eye disorders) | 0 | 1 | 0
Cholecystitis Infective (Infections and infestations) | 0 | 1 | 0
Corneal Erosion (Eye disorders) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Eyelid Cyst (Eye disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypertonic Bladder (Renal and urinary disorders) | 0 | 1 | 0
Iritis (Eye disorders) | 0 | 1 | 0
Pharyngitis Streptococcal (Infections and infestations) | 0 | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9 | 1/10 | 0/9
Renal Mass (Renal and urinary disorders) | 0 | 1 | 0
Retinal Degeneration (Eye disorders) | 0 | 1 | 0
Retinal Depigmentation (Eye disorders) | 0 | 1 | 0
Seasonal Allergy (Immune system disorders) | 0 | 1 | 0
Visual Impairment (Eye disorders) | 0 | 1 | 0
Vitreous Disorder (Eye disorders) | 0 | 1 | 0
Vitreous Opacities (Eye disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Conjunctival Granuloma (Eye disorders) | 0 | 0 | 1
Dry Eye (Eye disorders) | 0 | 0 | 1
Episcleritis (Eye disorders) | 0 | 0 | 1
Eyelid Ptosis (Eye disorders) | 0 | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 0 | 1
Macular Oedema (Eye disorders) | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Retinal Aneurysm (Eye disorders) | 0 | 0 | 1
Scleral Disorder (Eye disorders) | 0 | 0 | 1
Strabismus Correction (Surgical and medical procedures) | 0 | 0 | 1
Tooth Abscess (Infections and infestations) | 0 | 0 | 1
Tooth Infection (Infections and infestations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.